CLINICAL TRIAL: NCT05225350
Title: Matkassen-effekter av 3 månaders Intensiv Kostintervention Riktad Till Barn Med Fetma / Family Meals on Prescription- a Randomized Controlled Trial
Brief Title: Family Meals on Prescription- a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Region Halland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19002468
Record Dates: First submitted 2020-11-27; First posted 2022-02-04 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Childhood; Hypertension; Metabolic Syndrome; Dietary Habits
MeSH Terms: conditions — Pediatric Obesity; Hypertension; Metabolic Syndrome; Feeding Behavior | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Eligible children where randomized to 1 of 2 interventional arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (No Intervention): In the first arm the patients received care consistent with regional guidelines. Treatment as usual.
- Dietary Intervention (Experimental): In the second arm the patients received care consistent with regional guidelines in combination with the intensive dietary intervention for three months
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — See previous text
  Dietary intervention consisiting och each family recieving foodpackages for 5 dinner meals during three months.
  Arms: Dietary Intervention

SUMMARY:
"Matkassen - effekten av tre månaders intensiv kostintervention hos barn med fetma/ Family Meals on Prescription.- a randomized controlled trial : The aim of the study was to explore a novel approach for the treatment of obesity in children and adolescents through an intensive dietary intervention, consisting of receiving a weekly bag of groceries and recipes for five family meals at a reduced price for three months.

Data concerning dietary patterns and food habits, weight, BMI and blood markers for metabolic and cardiovascular disease was collected before the study began and again at the end of the study during the patients' one year follow up appointment at the clinics.

DETAILED DESCRIPTION:
Children between the age of 5-15 years receiving treatment for obesity at the pediatric clinics in Varberg and Kungsbacka were offered to participate in the trial.

The study population was divided into two arms including 60 patients in each arm:

* In the first arm the patients received care consistent with regional guidelines.
* In the second arm the patients received care consistent with regional guidelines in combination with the intensive dietary intervention for three months.

Data concerning dietary patterns and food habits, weight, BMI and blood markers for metabolic and cardiovascular disease was collected before the study began and again at the end of the study during the patients' one year follow up appointment at the clinics.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 5 to 15
* attending the Paediatric Obesity Clinics in Kungsbacka or Varberg

Exclusion Criteria:

* Younger than 5 or older than 15

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Dietary habits at one year | 1 year
  Assessment of meal pattern and dietary composition through questionaire.
Changes from Baseline in BMI at 3 months | 3 months
  Changes in BMI SDS in the different intervention groups
Changes from Baseline in BMI at 12 months | 12 months
  Changes in BMI SDS in the different intervention groups
Changes from Baseline in BMI at 18 months | 18 months
  Changes in BMI SDS in the different intervention groups
Changes from Baseline in BMI at 24 months | 24 months
  Changes in BMI SDS in the different intervention groups

SECONDARY OUTCOMES:
Changes from Baseline in metabolic parameters at 12 months | 12 months after treatment intervention
  Glucose control (fP-Glc, fs-Insulin, HbA1c,), Blood lipids (HDL, LDL, TG,), (liver function tests (, ALT, ) Vitamin D
Experience of intervention with in 1 year after intervention | with in 1 year after intervention
  Qualitative investigation through interviews and analysis from statements in medical journal

CONTACTS AND LOCATIONS:
Overall Officials: Lovisa Sjogren, MD, PhD, Principal Investigator — Goteborg University
Locations (1):
- Pediatric Clinic Region Halland, Halmstad, Halland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torstensson T, Almqvist-Tangen G, Waters S, Kindblom JM, Roswall J, Chaplin JE, Sjogren L. "The big win was that we actually cooked"- a qualitative interview study about the parental experience of Family Meals on Prescription for children living with obesity. J Health Popul Nutr. 2025 May 24;44(1):171. doi: 10.1186/s41043-025-00921-3. PMID 40413511
- [Derived] Torstensson T, Bohlin A, Almqvist-Tangen G, Roswall J, Kindblom JM, Sjogren L. Family meals on prescription as treatment for childhood obesity-a randomized controlled trial. Eur J Pediatr. 2024 Nov;183(11):4857-4866. doi: 10.1007/s00431-024-05744-8. Epub 2024 Sep 9. PMID 39251447